CLINICAL TRIAL: NCT05429164
Title: Comparison of the Effectiveness of Different Myofascial Release Techniques for the Pectoralis Minor Muscle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Büşra Aksan Sadıkoğlu, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IstanbulUC-2022
Record Dates: First submitted 2022-06-14; First posted 2022-06-23 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Pectoralis Minor Muscle Tension; Muscle Shortness; Mobility Limitation; Forward Scapular Posture; Rounded Shoulder Posture
MeSH Terms: conditions — Mobility Limitation | interventions — Myofascial Release Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Self Myofascial Release (Active Comparator): Self Myofascial Release only
  Interventions: Other: Self Myofascial Release
- Myofascial Release (Active Comparator): Myofascial Release with Physical Therapist Only
  Interventions: Other: Myofascial Release
- Instrument Assisted Soft Tissue Mobilization (Active Comparator): Instrument Assisted Soft Tissue Mobilization Only
  Interventions: Other: Instrument Assisted Soft Tissue Mobilization

INTERVENTIONS:
Other: Self Myofascial Release — In the self-myofascial release technique, a tennis ball will be placed on the 4th rib on the shoulder side to be applied on the wall, and the participants will be asked to move the ball using their body along the pectoralis minor.
  Arms: Self Myofascial Release
Other: Myofascial Release — A slight caudal force will be applied by the physiotherapist until the pectoralis minor muscle meets the comfortable elastic limit of the soft tissue.
  Arms: Myofascial Release
Other: Instrument Assisted Soft Tissue Mobilization — Instrument-assisted soft tissue mobilization will be performed with the specified instruments for the pectoralis minor muscle.
  Arms: Instrument Assisted Soft Tissue Mobilization

SUMMARY:
The aim of this study was to compare the effects of self-myofascial release, myofascial release with a physiotherapist and instrument assisted soft tissue mobilization (IASTM) techniques for the pectoralis minor muscle on pectoralis minor muscle length, rounded shoulder posture, glenohumeral joint total rotation range of motion (ROM) and skin temperature in asymptomatic individuals.

DETAILED DESCRIPTION:
In the literature, the effects of myofascial release and instrument assisted soft tissue mobilization (IASTM) applications on individuals with pectoralis minor muscle are investigated, but the available evidence is insufficient. In a study conducted in asymptomatic individuals, self-myofascial release was found to be more effective than placebo application in increasing glenohumeral flexion joint range of motion (ROM), improving pectoralis minor length and advanced scapular posture. However, there was one study comparing the short-term effectiveness of the self-myofascial release method and IASTM methods on pectoralis minor length, glenohumeral total arch movement and skin temperature in individuals with short pectoralis minor, and the results of both applications were found to be similar. Despite these studies in the current literature, the amount of evidence examining the effectiveness of myofascial release technique performed under the guidance of a physiotherapist in individuals with short pectoralis minor is insufficient. However, the number of studies comparing the immediate and short-term effects of different myofascial release methods on the pectoralis minor muscle lengthening is few. Given the limited evidence available, different myofascial release methods may produce different short-term responses on the pectoralis minor muscle, with different results on muscle length, scapular position, glenohumeral total arch motion, and superficial skin temperature. Therefore, the aim of this study was to compare the effects of 3 different myofascial release techniques on pectoralis minor muscle length, rounded shoulder posture, glenohumeral joint total rotation ROM and skin temperature in asymptomatic individuals.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 18-35
* Presence of pectoralis minor shortness
* Not having any upper extremity injury in the last 6 months

Exclusion Criteria:

* Presence of upper extremity surgery in the last 12 months
* Presence of neurological disorder in the upper extremity
* Any sensory problems or open wounds around the shoulder

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
pectoralis minor length | Baseline (first assessment)
  The length of the pectoralis minor muscle will be evaluated by the physiotherapist by calculating the pectoralis minor index (PMI), which is an objective evaluation method. In the calculation of PMI, the distance between the inferomedial of the coracoid process and the caudal edge of the 4th rib in the sternum will be evaluated with a tape measure to measure the length of the pectoralis minor muscle, and the values will be recorded in centimeters. Then, the measured pectoralis minor muscle length value will be calculated by dividing the participant's height in centimeters multiplied by 100. The reference value for PMI is 7.44%.

SECONDARY OUTCOMES:
pectoralis minor length | Immediately after the intervention (second assessment)
  The length of the pectoralis minor muscle will be evaluated by the physiotherapist by calculating the pectoralis minor index (PMI), which is an objective evaluation method. In the calculation of PMI, the distance between the inferomedial of the coracoid process and the caudal edge of the 4th rib in the sternum will be evaluated with a tape measure to measure the length of the pectoralis minor muscle, and the values will be recorded in centimeters. Then, the measured pectoralis minor muscle length value will be calculated by dividing the participant's height in centimeters multiplied by 100. The reference value for PMI is 7.44%.
rounded shoulder posture | Baseline (first assessment)
  The distance between the posterior border of the acromion and the table will be measured using a ruler while the patient is lying on her back, and the values will be recorded in cm
rounded shoulder posture | Immediately after the intervention (second assessment)
  The distance between the posterior border of the acromion and the table will be measured using a ruler while the patient is lying on her back, and the values will be recorded in cm.
glenohumeral joint total rotation ROM | Baseline (first assessment)
  The total value of the internal and external rotation angles of the glenohumeral joint will be measured with a digital inclinometer. After the inclinometer is placed on the patient's forearm, the glenohumeral joint total ROM will be recorded by passively externally and internally rotating the arms in the 90° flexion-90° abduction position.
glenohumeral joint total rotation ROM | Immediately after the intervention (second assessment)
  The total value of the internal and external rotation angles of the glenohumeral joint will be measured with a digital inclinometer. After the inclinometer is placed on the patient's forearm, the glenohumeral joint total ROM will be recorded by passively externally and internally rotating the arms in the 90° flexion-90° abduction position.
skin temperature | Baseline (first assessment)
  An infrared skin thermometer will be used to measure skin temperature.
skin temperature | Immediately after the intervention (second assessment)
  An infrared skin thermometer will be used to measure skin temperature.
number of trigger points | Baseline (first assessment)
  The presence of myofascial trigger points in the pectoralis minor muscle will be evaluated manually according to the Travel and Simons criteria. The total number will be recorded.
number of trigger points | Immediately after the intervention (second assessment)
  The presence of myofascial trigger point (MTN) in the pectoralis minor muscle will be evaluated manually according to the Travel and Simons criteria. The total number will be recorded.
pressure pain threshold | Baseline (first assessment)
  In order to evaluate the pain threshold of the pectoralis minor muscle, a pressure algometer (Baseline Push-Pull Force Gauge®, Fabrication Enterprises, Inc.) that can measure the pressure in pounds (Lb) and kilograms (kg), with a 1 cm diameter circular rubber disc attached to the piston at the end, will be used. Measurements will be recorded in kg/cm².
pressure pain threshold | Immediately after the intervention (second assessment)
  In order to evaluate the pain threshold of the pectoralis minor muscle, a pressure algometer (Baseline Push-Pull Force Gauge®, Fabrication Enterprises, Inc.) that can measure the pressure in pounds (Lb) and kilograms (kg), with a 1 cm diameter circular rubber disc attached to the piston at the end, will be used. Measurements will be recorded in kg/cm².

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided